CLINICAL TRIAL: NCT07206121
Title: A Feasibility Study for the SIRA-1000, SIRA® RFA Electrosurgical Device as an Adjunct to Breast Conserving Surgery
Brief Title: Feasibility Study for the SIRA-1000, SIRA® RFA Electrosurgical Device as an Adjunct to Breast Conserving Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innoblative Designs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 28001-CSP
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast-conserving Surgery; Breast Cancer - Infiltrating Ductal Carcinoma; ER/PR+Her2neu; Grade I, II, III
Keywords: Breast conserving surgery for breast cancer.
MeSH Terms: conditions — Breast Neoplasms; Lymphoma, Follicular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Safety study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Feasibility and safety study for women undergoing BCS. (Experimental): RFA electrosurgical device as an adjunct to BCS.
  Interventions: Device: Radiofrequency ablation alone; Device: Radiofrequency ablation Electrosurgical Device

INTERVENTIONS:
Device: Radiofrequency ablation alone — Demonstrate the accuracy of the device to produce approximately 1 cm depth of ablation around the tumor bed, as evaluated by post-ablation tissue samples at least 1cm deep.
Device: Radiofrequency ablation Electrosurgical Device — SIRA-1000 an radiofrequency ablation device, is designed to fit the post-lumpectomy cavity to provide uniform ablation.

SUMMARY:
This study aims to assess the safety and clinical accuracy of the SIRA-1000, SIRA® RFA Electrosurgical Device in ablating margins post-lumpectomy in patients undergoing breast conserving surgery for breast cancer. Radiofrequency ablation, or RFA, uses radio waves to create heat, that in turn, causes deliberate controlled damage to the tissue surrounding where the tumor was located. You may hear your doctor refer to this as the 'margins'. Your doctor is using this treatment to help destroy remaining cancer cells in the margins around the site of the lump.

DETAILED DESCRIPTION:
During your surgery, after your lump is removed, the surgeon will place the SIRA-1000 in the breast cavity and perform the RF ablation procedure to treat the margins of the lumpectomy surgical site. A stitch will be used to stabilize and secure the tissue around the neck of the SIRA-1000 to ensure that contact is maintained between the SIRA-1000 electrode array and cavity tissue.

Upon completion of the RF ablation treatment, your tumor and the tissue samples from the ablated edges of the surgical site will be sent for review under a microscope (pathology).

After this, your surgery will be completed as standard, and your discharge will be determined by your medical team like any other surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Biologic female
2. 50 years of age and older
3. Confirmed diagnosis of breast cancer:

   1. Infiltrating ductal carcinoma
   2. ER/PR+Her2neu-
   3. Grade I, II, or III
4. Unicentric, unilateral tumor size ≤ 3cm
5. Tumor location ≥ 2 cm from skin and other structures
6. Zubrod Performance Status of 0, 1, or 2
7. No palpable lymphadenopathy
8. Able and willing to provide written informed consent

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Neoadjuvant chemotherapy
3. Cardiac arrhythmia
4. Patients with active implantable medical devices, such as implanted cardiac pacemakers or defibrillators, or any other electronic device
5. Current or history of breast implants
6. Multi-centric or bilateral breast cancer
7. Diffuse microcalcifications
8. Participating in another ongoing clinical study in which concomitant diagnostic or therapeutic intervention that would reasonably be expected to alter the outcomes under study
9. Has a condition or is in a situation which in the Investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-02-06 (Estimated); Study Completion 2032-02-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of SIRA-1000 by summarizing the occurrence of Adverse Events. | The study will span a total of approximately 12 months with a follow-up for 5 years.
  Assess the occurrence adverse events and to evaluate the impact of RFA on healing process.
Healing Process assessed by BREAST-Q Questionnaire | 6 months
  Assess healing process using cosmesis and quality of life patient reported outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, MD, PhD, MSCHT, MAMSE, FACS, Study Chair
Locations (1):
- University of Texas Medical Branch at Galveston, TX, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study.

REFERENCES:
- [Background] Klimberg VS, Ochoa D, Henry-Tillman R, Hardee M, Boneti C, Adkins LL, McCarthy M, Tummel E, Lee J, Malak S, Makhoul I, Korourian S. Long-term results of phase II ablation after breast lumpectomy added to extend intraoperative margins (ABLATE l) trial. J Am Coll Surg. 2014 Apr;218(4):741-9. doi: 10.1016/j.jamcollsurg.2013.12.032. Epub 2014 Jan 11. PMID 24655863
- See also: Innoblative Designs, Inc. website — https://innoblative.com/